CLINICAL TRIAL: NCT04857281
Title: Non-invasive Vagal Nerve Stimulation (nVNS) for Symptomatic Exacerbation of Nausea in Patients With Gastroparesis and Related Disorders
Acronym: nVNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00265410
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Unexplained Nausea and Vomiting; Gastroparesis
MeSH Terms: conditions — Vomiting; Gastroparesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- nVNS device (Experimental): Candidates who, after the screening period are eligible to receive the nVNS device.
  Interventions: Device: nVNS (gammaCore)

INTERVENTIONS:
Device: nVNS (gammaCore) — The treatment will be self-administered using nVNS and will be applied for 4 weeks; a member of the study will provide the proper training on the correct use of nVNS. The patient will be instructed to use the nVNS in place of the rescue medications. When the nauseas gets bad enough that they feel to use a rescue medication they will first use the device on one side of the neck for two 2-minute stimulations and wait fifteen minutes to check if the stimulation works. If this does not help either, they will stimulate with an additional 2 stimulations and wait for another fifteen minutes. If there is no improvement rescue medication will be used. nVNS can be used up to, but no more than, 8 times a day.

SUMMARY:
The hypothesis of this pilot study is that nVNS will result in relief of nausea by modulation of vagal nerve activity. nVNS is the first non-invasive, handheld medical device applied on the side of the neck and sends gentle, patented mild electrical stimulation through the skin to activate the vagus nerve. nVNS offers a potential alternative to Gastric electrical stimulation (GES) that could eliminate significant risks of injury or illness or identify likely responders to implantable neurostimulator including implanted VNS (iVNS). nVNS could provide a more effective and safer alternative to the use of traditional rescue medications.

DETAILED DESCRIPTION:
The patient will receive the gammaCore (nVNS) device and a video instruction will be use to explain how to properly handle the device. Treatment can only start after eligibility has been fully checked and all data collected at screening have been keyed into the trial database.

The patient will be instructed to use the nVNS in place of the rescue medications. When the nauseas gets bad enough that they feel to use a rescue medication they will first use the device on one side of the neck for two 2-minute stimulations and wait fifteen minutes to check if the stimulation works. If this does not help either, they will stimulate with an additional 2 stimulations and wait for another fifteen minutes. If there is no improvement rescue medication will be used. nVNS can be used up to, but no more than, 8 times a day.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at registration.
* Diagnosis of gastroparesis as documented by gastric emptying scintigraphy (4-hour emptying after a low-fat meal with any combination of 2- and 4-hour retention of >60% and 10%, respectively), or Chronic Unexplained Nausea and Vomiting (CUNV).
* Ongoing symptoms (i.e. Nausea and vomiting, bloating, and abdominal pain) with a nausea score of 3 or more on the patient assessment of upper gastrointestinal disorders-symptom severity index (PAGI-SYM) scale at baseline (moderate to severe nausea).
* Exclusion of other causes of symptoms such as mechanical gastrointestinal obstruction, uncontrolled esophagitis, peptic ulcer disease, etc. By standard radiographic or endoscopic tests.
* Use of the following medications on an as-needed basis: ondansetron, promethazine or prochlorperazine but no more than four times a day.

Exclusion Criteria:

* Another active disorder, which could explain symptoms in the opinion of the investigator.
* Age < than 18 years.
* Pregnancy or nursing.
* A previous surgery of the upper gastrointestinal tract, including vagotomy.
* Use of narcotics more than 3 days per week.
* History of prolonged QT interval or a history of clinically significant arrhythmia.
* Abnormal baseline ECG (e.g. Second- and third-degree heart block, atrial fibrillation, atrial flutter, recent history of ventricular tachycardia or ventricular fibrillation, or clinically significant premature ventricular contraction).
* Previous bilateral or right cervical vagotomy.
* Uncontrolled high blood pressure.
* Currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
* History of carotid endarterectomy or vascular neck surgery on the right side.
* Implanted with metal cervical spine hardware or has a metallic implant near the gammaCore stimulation site.
* Any other condition, which in the opinion of the investigator would impede compliance or hinder the completion of the study.
* Failure to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pasricha, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barahona G, de Barahona LV, Sidhu SS, Burns R, McKnight M, Hui KY, Bulat R, Treisman GJ, Liebler E, McClure CK, Pasricha PJ. Non-invasive Vagal Nerve Stimulation Decreases the Need for Rescue Medication for Nausea Exacerbation in Patients with Chronic Nausea and Vomiting. Dig Dis Sci. 2025 Oct 16. doi: 10.1007/s10620-025-09457-2. Online ahead of print. PMID 41100038

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After meeting the criteria, patients underwent a 7-day screening to establish baseline symptoms and nausea medication intake. Subjects were then randomly assigned to use the nVNS device on one side of the neck for 4 weeks. This was followed by a 2-week washout period before switching to the opposite side, with an additional 2-week washout at the end.
Groups:
- nVNS Was First Applied to One Side of the Neck, Followed by Stimulation on the Opposite Side.: After meeting the criteria, patients underwent a 7-day screening to establish baseline symptoms and nausea medication intake. Candidates who were eligible after the screening were then randomly assigned to use the nVNS (gammaCore) device on one side of the neck for 4 weeks, followed by a 2-week washout period before switching to the opposite side, with an additional 2-week washout at the end. Eight subjects were excluded before starting nVNS due to missing baseline information on symptoms and nausea medication intake.
  The treatment with nVNS will be self-administered for 4 weeks, with proper training provided by a study member on the correct use of the device. Patients will be instructed to use nVNS instead of rescue medications. When nausea becomes severe, patients will first apply two 2-minute stimulations on one side of the neck and wait 15 minutes to assess its effectiveness. If the nausea persists, they will apply an additional two stimulations and wait another 15 minutes. If there is still no improvement, they may use rescue medication. nVNS can be used up to 8 times per day, but no more.
Period: Baseline
Arm/Group | nVNS Was First Applied to One Side of the Neck, Followed by Stimulation on the Opposite Side.
Started | 49
Completed | 41
Not Completed | 8
Period: First Intervention - 4 Weeks
Arm/Group | nVNS Was First Applied to One Side of the Neck, Followed by Stimulation on the Opposite Side.
Started | 41
Completed | 41
Not Completed | 0
Period: First Washout - 2 Weeks
Arm/Group | nVNS Was First Applied to One Side of the Neck, Followed by Stimulation on the Opposite Side.
Started | 41
Completed | 41
Not Completed | 0
Period: Second Intervention - 4 Weeks
Arm/Group | nVNS Was First Applied to One Side of the Neck, Followed by Stimulation on the Opposite Side.
Started | 41
Completed | 41
Not Completed | 0
Period: Second Washout - 2 Weeks
Arm/Group | nVNS Was First Applied to One Side of the Neck, Followed by Stimulation on the Opposite Side.
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | nVNS Was First Applied to One Side of the Neck, Followed by Stimulation on the Opposite Side.
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 1
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 34 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Use of Rescue Medications for Exacerbation of Nausea/Vomiting.
Description: Average daily use of rescue medications for exacerbation of nausea/vomiting = sum of nausea medications / number of days with non-missing nausea medication data.
Time Frame: Baseline, 4, 6, 10 and 12 weeks of study participation
Population: The analysis included only participants who completed each study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: medications/day
Arm/Group | nVNS Was First Applied to One Side of the Neck, Followed by Stimulation on the Opposite Side.
Number analyzed (Participants) | 41
medications/day
  Baseline | 1.186 [0.675 to 1.696]
  First Side (4 Weeks Follow-up) | 0.551 [0.327 to 0.776]
  Wash Out (6 Weeks Follow-up) | 0.754 [0.439 to 1.070]
  Second Side (10 Weeks Follow-up) | 0.447 [0.221 to 0.673]
  Final Wash Out (12 Weeks Follow-up) | 0.537 [0.183 to 0.892]

ADVERSE EVENTS:
Time Frame: Up to 13 weeks
Description: Serious Adverse Events and All-cause mortality were not collected for any participant. Other not serious adverse events were not collected for eight subjects who were excluded before starting nVNS.
Arm/Group | nVNS Device
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 1/41
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | nVNS Device (N=41)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT04857281/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT04857281/ICF_001.pdf